CLINICAL TRIAL: NCT00995176
Title: The Women's HIV SeroIncidence Study (ISIS)
Status: Completed | Type: Observational
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HPTN 064; 1U01AI068619 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
Keywords: Prevention; HIV; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women residing in areas from defined geographic areas with high HIV prevalence and poverty
- 2: Men residing in areas from defined geographic areas with high HIV prevalence and poverty

SUMMARY:
Approximately 30 percent of new HIV infections in the Unites States occur in women, with a disproportionate number occurring in women of color. This observational study has been designed to help determine the HIV incidence among women in the study communities as well as to identify steps that women can take to lower their HIV-infection risk.

DETAILED DESCRIPTION:
In 1985 women accounted for only 8 percent of new AIDS diagnoses in the United States. Today women are estimated to account for nearly 30 percent of the people who are diagnosed with new HIV infections (incidence). A disproportionate amount of those infections (80 percent) occur among Black and Hispanic girls and women. This observational study has been designed to help determine the HIV incidence among women in the study communities as well as to identify steps that women can take to lower their HIV-infection risk.

Research teams will conduct eligibility screening interviews with women whom they have encountered in various locations within the study communities. Eligibility screenings, as well as subsequent study visits, will take place in a variety of mutually agreeable locations that are capable of providing both privacy and confidentiality. Examples include clinics, mobile vans, community organizations or other appropriate public places. The eligibility interview contains topics related to sexual behavior, drug and alcohol use, incarceration history and previous STI diagnosis and treatment. Information about where the potential participant resides and her current sexual partners will also be gathered.

The women who are found to be eligible will be asked to provide a blood sample for HIV and other investigational testing. They will also be asked to participate in a longer interview. All participants will receive HIV risk-reduction counseling, free condoms and appropriate referrals. Monthly contact will be maintained with participants through information that was provided upon enrollment. A phone number that participants can use to contact the research team will also be provided. Monthly calls will each last about 5 to 15 minutes.

About six months after enrolling each participant will be scheduled to have another in-person visit with study staff to complete an interview similar to the eligibility interview. Women who have tested HIV negative will be asked to provide another blood sample for HIV testing during that same period of time, while women who are living with HIV will be asked to provide blood samples to evaluate their HIV-related health. Women who enroll during the earliest portion of the study may be asked to complete a second visit in another six months. Those women will continue to receive monthly contacts between the dates of their first and second visits.

In addition to the primary participant group, a small group of women from four of the study communities will also be recruited to participate in interviews and focus groups that will cover issues similar to the topics included in the eligibly screening. A small group of men from those same four study communities will also be recruited to participate in similar focus groups.

ELIGIBILITY:
HPTN 064, potential participants will be approached at randomly selected locations within study communities. As a result, potential participants are not able to self-refer directly through phone, email or in-person.

Inclusion Criteria for Women:

* Self identify as a woman
* 18 to 44 years of age, inclusive on the date of screening
* Willing to receive HIV test results
* Resides in a designated study community
* Has engaged in unprotected (e.g. without a condom) vaginal and/or anal sex with a man during the prior 6 months
* At least one of the following criteria:

  * Illicit injected and/or noninjected drug use (e.g. heroin, cocaine, crack cocaine, methamphetamine, and/or prescription drugs used outside the oversight of a medical professional) within 6 months. Participants whose only illicit drug use is marijuana do not meet the illicit drug use eligibility criteria.
  * Alcohol dependence (within 6 months)
  * Binge drinking defined as four or more drinks at one time (e.g. during the morning, afternoon or evening) within 6 months
  * Incarceration within 5 years (jail and/or prison)
  * STI (gonorrhea, Chlamydia, trichomonas, or syphilis) within 6 months
  * Exchange of sex for commodities (e.g. drugs, money, shelter) within 6 months
  * Male sexual partner within 6 months with any history of self-reported use of illicit injected or noninjected drugs within 6 months, incarceration (within 5 years), STIs (within 6 months), HIV-infected diagnosis, or history of binge drinking defined as 5 or more drinks at one time (within 6 months) and/or alcohol dependence (within 6 months)

Inclusion Criteria for Men:

* Self identify as a man
* 18 years of age or older
* Resides in a designated community
* Unprotected vaginal and/or anal sex with a woman during the prior 6 months
* At least one of the following criteria:

  * Illicit injected and/or noninjected drug use within 6 months
  * Alcohol dependence (within 6 months)
  * Binge drinking defined as five or more drinks at one time (e.g. during the morning, afternoon or evening) within 6 months
  * Incarceration (within 5 years, including jail and/or prison)
  * STI within 6 months
  * Exchange of sex for commodities
  * HIV-infected

Exclusion Criteria for Women:

* History of prior HIV-infected diagnosis
* Planning on moving out of state within the study follow-up period or traveling out of state for more than 2 consecutive months during the study follow-up period
* Current enrollment in an HIV prevention trial
* Current or past participation in an HIV vaccine trial
* Any condition that, in the opinion of the study staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Exclusion Criteria for Men:

* Any condition that, in the opinion of the study staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women residing in areas from defined geographic areas with high HIV prevalence and poverty
Sampling Method: Probability Sample
Enrollment: 2099 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Estimation of the overall HIV-1 incidence rate among 2,000 women in the US from defined geographic areas with high HIV prevalence and poverty | Throughout study

SECONDARY OUTCOMES:
Evaluation of laboratory assays for HIV-1 incidence determination | Throughout study
Estimation of recruitment and retention rates | Throughout study
Assessment of women's preferred recruitment and retention strategies for future studies | Throughout study
Description of social, structural, and contextual factors in a subgroup of female participants to inform future intervention studies | Throughout study
Estimation of HIV-1 prevalence rate among women who have not reported previously testing HIV positive | Throughout study
Exploration of facilitators and barriers to HIV testing among men residing in high risk areas to inform future studies | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sally Hodder, MD, Study Chair — UMDNJ - New Jersey Medical School; Jessica Justman, Study Chair — Columbia University
Locations (9):
- United States (9):
  - George Washington University, Washington D.C., District of Columbia
  - The Ponce de Leon Center, Atlanta, Georgia
  - Hope Clinic of the Emory Vaccine Center, Decatur, Georgia
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Harlem Prevention Ctr. CRS, New York, New York
  - Bronx- Lebanon Hospital Center Clinical Research Site, The Bronx, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Wake County Health and Human Services, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
Data was collated into manuscripts by the statistical and data management center for the HPTN.

REFERENCES:
- [Background] Hodder SL, Justman J, Haley DF, Adimora AA, Fogel CI, Golin CE, O'Leary A, Soto-Torres L, Wingood G, El-Sadr WM; HIV Prevention Trials Network Domestic Prevention in Women Working Group. Challenges of a hidden epidemic: HIV prevention among women in the United States. J Acquir Immune Defic Syndr. 2010 Dec;55 Suppl 2(Suppl 2):S69-73. doi: 10.1097/QAI.0b013e3181fbbdf9. PMID 21406990
- [Background] Haley DF, Justman JE. The HIV epidemic among women in the United States: a persistent puzzle. J Womens Health (Larchmt). 2013 Sep;22(9):715-7. doi: 10.1089/jwh.2013.4562. No abstract available. PMID 24007379
- [Background] Haley DF, Lucas J, Golin CE, Wang J, Hughes JP, Emel L, El-Sadr W, Frew PM, Justman J, Adimora AA, Watson CC, Mannheimer S, Rompalo A, Soto-Torres L, Tims-Cook Z, Carter Y, Hodder SL; HPTN 064 Study Team. Retention strategies and factors associated with missed visits among low income women at increased risk of HIV acquisition in the US (HPTN 064). AIDS Patient Care STDS. 2014 Apr;28(4):206-17. doi: 10.1089/apc.2013.0366. PMID 24697160
- [Result] Eshleman SH, Hughes JP, Laeyendecker O, Wang J, Brookmeyer R, Johnson-Lewis L, Mullis CE, Hackett J Jr, Vallari AS, Justman J, Hodder S. Use of a multifaceted approach to analyze HIV incidence in a cohort study of women in the United States: HIV Prevention Trials Network 064 Study. J Infect Dis. 2013 Jan 15;207(2):223-31. doi: 10.1093/infdis/jis658. Epub 2012 Nov 5. PMID 23129758
- [Result] Hodder SL, Justman J, Hughes JP, Wang J, Haley DF, Adimora AA, Del Rio C, Golin CE, Kuo I, Rompalo A, Soto-Torres L, Mannheimer SB, Johnson-Lewis L, Eshleman SH, El-Sadr WM; HIV Prevention Trials Network 064; Women's HIV SeroIncidence Study Team. HIV acquisition among women from selected areas of the United States: a cohort study. Ann Intern Med. 2013 Jan 1;158(1):10-8. doi: 10.7326/0003-4819-158-1-201301010-00004. PMID 23277896
- [Result] Adimora AA, Hughes JP, Wang J, Haley DF, Golin CE, Magnus M, Rompalo A, Justman J, del Rio C, El-Sadr W, Mannheimer S, Soto-Torres L, Hodder SL; HPTN 064 Protocol Team. Characteristics of multiple and concurrent partnerships among women at high risk for HIV infection. J Acquir Immune Defic Syndr. 2014 Jan 1;65(1):99-106. doi: 10.1097/QAI.0b013e3182a9c22a. PMID 24056163
- [Result] Haley DF, Golin C, El-Sadr W, Hughes JP, Wang J, Roman Isler M, Mannheimer S, Kuo I, Lucas J, DiNenno E, Justman J, Frew PM, Emel L, Rompalo A, Polk S, Adimora AA, Rodriquez L, Soto-Torres L, Hodder S. Venue-based recruitment of women at elevated risk for HIV: an HIV Prevention Trials Network study. J Womens Health (Larchmt). 2014 Jun;23(6):541-51. doi: 10.1089/jwh.2013.4654. Epub 2014 Apr 17. PMID 24742266
- [Result] Kuo I, Golin CE, Wang J, Haley DF, Hughes J, Mannheimer S, Justman J, Rompalo A, Frew PM, Adimora AA, Soto-Torres L, Hodder S; HPTN 064 Study Team. Substance use patterns and factors associated with changes over time in a cohort of heterosexual women at risk for HIV acquisition in the United States. Drug Alcohol Depend. 2014 Jun 1;139:93-9. doi: 10.1016/j.drugalcdep.2014.03.007. Epub 2014 Mar 19. PMID 24698079
- [Derived] Abrams JA, Odlum M, Tillett E, Haley D, Justman J, Hodder S, Vo L, O'Leary A, Frew PM; HIV Prevention Trials Network 064 (HTPN) Study Team. Strategies for increasing impact, engagement, and accessibility in HIV prevention programs: suggestions from women in urban high HIV burden counties in the Eastern United States (HPTN 064). BMC Public Health. 2020 Sep 3;20(1):1340. doi: 10.1186/s12889-020-09426-6. PMID 32883248
- [Derived] Frew PM, Parker K, Vo L, Haley D, O'Leary A, Diallo DD, Golin CE, Kuo I, Soto-Torres L, Wang J, Adimora AA, Randall LA, Del Rio C, Hodder S; HIV Prevention Trials Network 064 (HTPN) Study Team. Socioecological factors influencing women's HIV risk in the United States: qualitative findings from the women's HIV SeroIncidence study (HPTN 064). BMC Public Health. 2016 Aug 17;16(1):803. doi: 10.1186/s12889-016-3364-7. PMID 27530401